CLINICAL TRIAL: NCT02461212
Title: Validation of HepaFat-Scan for Noninvasive Measurement of Steatosis in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Resonance Health (Industry)
Responsible Party: Principal Investigator, Miriam Vos, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00078470
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: HepaFat-Scan; Liver Disease; Pediatrics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liver MRI (Experimental): Liver MRI imaging will be performed on subjects undergoing a liver biopsy
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)
- Liver MRI repositioned (Experimental): Liver MRI imaging will be performed on subjects undergoing a liver biopsy and then they will be repositioned and will repeat the MRI
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — A MRI scan which will include magnetic resonance spectroscopy (MRS) of the liver to determine hepatic triglyceride content, a hepafat scan to measure volume fraction of fat in liver tissue, and a MRI for detection of liver fibrosis. The scan will last approximately 15 minutes.

SUMMARY:
The purpose of this study is to see if the HepaFat-Scan (a special sequence of images done in a MRI) can accurately detect the amount of fat in the liver.

DETAILED DESCRIPTION:
The leading cause of liver disease for both adults and children in the US is nonalcoholic fatty liver disease (NAFLD), an obesity-related liver disease closely associated with the metabolic syndrome. NAFLD increases the risk of liver disease but also increases risk of type II diabetes, cardiovascular disease (CVD) and the metabolic syndrome. Invasive liver biopsy has been considered the best diagnostic tool for confirming NAFLD. This study will establish magnetic resonance imaging (MRI) / magnetic resonance spectroscopy (MRS) as a quantitative noninvasive "virtual biopsy" and benefit the health of children with liver diseases by decreasing risk and improving diagnosis. Specifically, in NAFLD, this fat quantification protocol will be broadly useful in future research studies, including therapies for NAFLD as well as for patient diagnosis and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls age 7-18 years
* Scheduled for a clinically indicated liver biopsy
* Able to undergo MRI without sedation
* Written informed consent from parent or legal guardian
* Written informed assent from the child when indicated by age

Exclusion Criteria:

* Renal disease with a creatinine > 2 or requiring dialysis
* Metal, braces or other implanted devices not compatible with MRI
* Not willing to try to hold still for an un-sedated MRI
* Pregnancy
* Failure to give consent or assent

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Correlation between HepaFat-Scan and pathology based assessment of steatosis | 12 months
  Correlation of histologic steatosis to HepaFat-Scan measurement.
Correlation of HepaFat-Scan measurement with magnetic resonance spectroscopy (MRS) and computerized steatosis | 12 months
  The percent of total steatosis by MRS and computerized steatosis (computer-assisted pixel count algorithm) will be plotted and Pearson correlation coefficient will be calculated to explore their relationship.
Correlation of HepaFat-Scan measurement with magnetic resonance spectroscopy (MRS) and grade of pathology of assessment | 12 months
  The percent steatosis from the MRS and grade of pathology of assessment will be plotted and compared to categorization using HepaFat-Scan.
Repeatability of HepaFat-Scan | 12 months
  Two HepaFat-Scans will be done on half of the subjects. Repeatability of the Hepafat scan will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam B Vos, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States